CLINICAL TRIAL: NCT00002515
Title: Myeloablative Chemotherapy With Bone Marrow Rescue For Rare Poor-Prognosis Cancers
Brief Title: Combination Chemotherapy Followed by Bone Marrow Transplantation in Treating Patients With Rare Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Purpose: Treatment
Other Study IDs: 92-148; CDR0000078115 (Registry Identifier: PDQ (Physician Data Query)); NCI-V93-0214
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-06

CONDITIONS: Childhood Germ Cell Tumor; Extragonadal Germ Cell Tumor; Head and Neck Cancer; Kidney Cancer; Liver Cancer; Lymphoma; Neuroblastoma; Ovarian Cancer; Retinoblastoma; Sarcoma; Testicular Germ Cell Tumor
Keywords: chondrosarcoma; recurrent childhood rhabdomyosarcoma; stage IV childhood liver cancer; recurrent neuroblastoma; recurrent childhood liver cancer; recurrent Wilms tumor and other childhood kidney tumors; stage IV Wilms tumor; recurrent retinoblastoma; stage IV childhood lymphoblastic lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent osteosarcoma; stage IV ovarian germ cell tumor; recurrent malignant testicular germ cell tumor; childhood germ cell tumor; alveolar childhood rhabdomyosarcoma; recurrent childhood soft tissue sarcoma; recurrent ovarian germ cell tumor; childhood fibrosarcoma; extragonadal germ cell tumor; childhood desmoplastic small round cell tumor; recurrent childhood small noncleaved cell lymphoma; stage IV childhood small noncleaved cell lymphoma; recurrent childhood large cell lymphoma; stage IV childhood large cell lymphoma; recurrent Ewing sarcoma/peripheral primitive neuroectodermal tumor; stage IV lymphoepithelioma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; recurrent lymphoepithelioma of the nasopharynx
MeSH Terms: conditions — Head and Neck Neoplasms; Kidney Neoplasms; Liver Neoplasms; Lymphoma; Neuroblastoma; Ovarian Neoplasms; Retinoblastoma; Sarcoma; Testicular Germ Cell Tumor; Chondrosarcoma; Wilms Tumor; Osteosarcoma; Testicular Neoplasms; Fibrosarcoma; Desmoplastic Small Round Cell Tumor; Burkitt Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Neuroectodermal Tumors, Primitive, Peripheral | interventions — Filgrastim; Carboplatin; Thiotepa; Topotecan

INTERVENTIONS:
Biological: filgrastim
Drug: carboplatin
Drug: thiotepa
Drug: topotecan hydrochloride
Procedure: autologous bone marrow transplantation
Procedure: bone marrow ablation with stem cell support
Procedure: in vitro-treated bone marrow transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Bone marrow transplantation may allow doctors to give higher doses of chemotherapy and kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy with thiotepa, carboplatin, and topotecan followed by bone marrow transplantation in treating patients who have metastatic or progressive rare cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Improve the long term disease-free survival of patients with rare cancers at high risk for lethal relapse by using myeloablative chemotherapy with thiotepa, carboplatin, and topotecan followed by autologous bone marrow or peripheral blood stem cell rescue.

OUTLINE: Autologous bone marrow or peripheral blood stem cells (PBSC) are harvested. Patients receive high-dose thiotepa IV over 3 hours on days -8 to -6, carboplatin IV over 4 hours on days -5 to -3, and topotecan IV over 30 minutes on days -8 to -4. Autologous bone marrow or PBSC are reinfused on day 0. Patients receive filgrastim (G-CSF) IV twice daily beginning on day 1.

Patients are followed for 1 year.

PROJECTED ACCRUAL: Approximately 50 patients will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignancy of one of the following types:

  * Wilms' tumor
  * Liver cancer
  * Desmoplastic or other small round cell tumor
  * Nasopharyngeal carcinoma
  * Fibrosarcoma
* Disease that has metastasized and has a cure rate of no greater than 25% with conventional treatment or disease that has progressed after prior chemotherapy, was not then surgically resectable, and has a salvage rate with nonmyeloablative therapies of no greater than 25% required
* Maximal benefit from conventional (nonmyeloablative) doses of combination chemotherapy required prior to entry, and it is recommended that patients have received a minimum of one of the following:

  * 2 courses of high-dose cyclophosphamide (as per protocol MSKCC-90062)
  * 2 courses of high-dose ifosfamide/etoposide (as in the poor-risk sarcoma protocol MSKCC-90071A)
  * 1 course of high-dose cyclophosphamide plus 1 course of high-dose ifosfamide/etoposide
* Within 3 weeks of initiation of protocol therapy, patients must be:

  * In CR or good PR OR
  * Tumor considered "chemosensitive", i.e., a 50% or greater decrease in at least 1 measurable tumor parameter attributable to prior chemotherapy without evidence of progressive disease by any other parameter
* Ineligible for other IRB-approved myeloablative regimens
* No evidence of current bone marrow involvement on bone marrow aspiration (x4) and biopsy (x2)

PATIENT CHARACTERISTICS:

Age:

* 21 and under

Performance status:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT no greater than 1.5 times ULN
* Alkaline phosphatase no greater than 1.5 times ULN
* 5'-Nucleotidase no greater than 1.5 times ULN

Renal:

* Creatinine normal
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* CPK normal
* Echocardiogram (or RNCA) normal
* EKG normal

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* See Disease Characteristics

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 1992-10; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian H. Kushner, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States